CLINICAL TRIAL: NCT04771715
Title: An Observational Real-world Study of Regorafenib Plus Programmed Cell Death-1 (PD-1) Inhibitors in Chinese Patients With Advanced Colorectal Cancer
Brief Title: Regorafenib Plus Programmed Cell Death-1 (PD-1) Inhibitors in Patients With Advanced Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S-K1517
Record Dates: First submitted 2021-02-17; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Advanced Colorectal Carcinoma
MeSH Terms: interventions — regorafenib; Nivolumab; pembrolizumab; camrelizumab; sintilimab; toripalimab; tislelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Regorafenib — Medical records are reviewed to identify participants who received at least one dose of regorafenib plus a PD-1 inhibitor (nivolumab/pembrolizumab/camrelizumab/sintilimab/toripalimab/tislelizumab) in routine medical care.
  Other Names: Stivarga
Drug: Nivolumab — Medical records are reviewed to identify participants who received at least one dose of regorafenib plus a PD-1 inhibitor (nivolumab/pembrolizumab/camrelizumab/sintilimab/toripalimab/tislelizumab) in routine medical care.
  Other Names: Opdivo
Drug: Pembrolizumab — Medical records are reviewed to identify participants who received at least one dose of regorafenib plus a PD-1 inhibitor (nivolumab/pembrolizumab/camrelizumab/sintilimab/toripalimab/tislelizumab) in routine medical care.
  Other Names: Keytruda
Drug: Camrelizumab — Medical records are reviewed to identify participants who received at least one dose of regorafenib plus a PD-1 inhibitor (nivolumab/pembrolizumab/camrelizumab/sintilimab/toripalimab/tislelizumab) in routine medical care.
Drug: Sintilimab — Medical records are reviewed to identify participants who received at least one dose of regorafenib plus a PD-1 inhibitor (nivolumab/pembrolizumab/camrelizumab/sintilimab/toripalimab/tislelizumab) in routine medical care.
Drug: Toripalimab — Medical records are reviewed to identify participants who received at least one dose of regorafenib plus a PD-1 inhibitor (nivolumab/pembrolizumab/camrelizumab/sintilimab/toripalimab/tislelizumab) in routine medical care.
Drug: Tislelizumab — Medical records are reviewed to identify participants who received at least one dose of regorafenib plus a PD-1 inhibitor (nivolumab/pembrolizumab/camrelizumab/sintilimab/toripalimab/tislelizumab) in routine medical care.

SUMMARY:
This is a multicenter observational study aimed to describe the efficacy and safety of regorafenib plus programmed cell death-1 (PD-1) inhibitors in Chinese patients with advanced colorectal cancer in routine clinical practice. The primary end point is overall survival. The secondary endpoints include progression-free survival, objective response rate, disease control rate and the incidence of treatment-related adverse events.

DETAILED DESCRIPTION:
The investigators retrospectively identify patients with advanced colorectal adenocarcinoma who received at least one dose of PD-1 inhibitors plus regorafenib from 5/2019 to 2/2021 in 14 Chinese medical centers. Patients received the study treatment as part of routine medical care based on the consensus of clinicians and patients. In addition to the primary and secondary outcomes, other patient and treatment characteristics including baseline microsatellite instability status, metastatic sites, previous treatment regimens, post-treatment regimens, are collected in order to describe the real-world treatment patterns.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Histologically or cytologically confirmed advanced or metastatic colorectal adenocarcinoma
3. Disease progression on standard of care therapy
4. Patients must have received at least one dose of PD-1 inhibitors in combination with regorafenib
5. At least one available laboratory or vital sign measurement obtained subsequent to at least one dose of study treatment for safety analysis
6. Confirmed treatment discontinuation/disease progression/available radiological evaluation or at least eight weeks of follow-up subsequent to the first dose of study treatment for efficacy analysis
7. Prior exposure to regorafenib monotherapy or a PD-1 inhibitor monotherapy was allowed

Exclusion Criteria:

1. Other malignancies within the past 5 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinoma of the skin
2. Participation in other interventional studies while receiving regorafenib plus a PD-1 inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators performed a retrospective review of medical records to identify patients with advanced colorectal cancer who received at least one dose of PD-1 inhibitors in combination with regorafenib as routine medical care in 14 Chinese medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 24 months
  The time from treatment initiation to death due to any cause

SECONDARY OUTCOMES:
Progression-free survival | Up to 24 months
  The time from treatment initiation to the first documented disease progression or death due to any cause, whichever occurs first
Objective response rate (ORR) | Up to 12 months
  The proportion of participants in the analysis population who have complete response (CR) or partial response (PR) determined by investigators using RECIST 1.1 criteria at any time during the study
Disease control rate (DCR) | Up to 12 months
  The proportion of participants in the analysis population who have CR, PR or stable disease (SD) determined by investigators using RECIST 1.1 criteria at any time during the study
Incidence of treatment-related adverse events (TRAE) | Up to 24 months
  Percentage of participants with TRAEs as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang K, Han L, Wu S, Qu X, Li Q, Zhao C, Zhou J, Jin X, Wang Y, Yan D, Cheng Z, Hua Y, Zhang Y, Ge Y, Sun J, Deng W, Zhao L, Zhao Y. Real-world outcomes of regorafenib combined with immune checkpoint inhibitors in patients with advanced or metastatic microsatellite stable colorectal cancer: A multicenter study. Cancer Immunol Immunother. 2022 Jun;71(6):1443-1451. doi: 10.1007/s00262-021-03083-3. Epub 2021 Oct 24. PMID 34689233